CLINICAL TRIAL: NCT03367247
Title: BOLSTER: Building Out Lifelines for Safety, Trust, Empowerment and Renewal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alexi A. Wright, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 17-475; CA166210 (Other: NCI); R21CA223684 (NIH)
Record Dates: First submitted 2017-11-28; First posted 2017-12-08 (Actual); Results first posted 2023-08-15 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Gynecologic Cancer; Gastrointestinal Cancer
Keywords: Ovarian Cancer; Bowel blockage; Ascites; Supportive care; Nursing; Mobile health; m-Health; Tele-health; Palliative Care; Symptom management; Gastrointestinal Cancer; Gynecologic Cancer; Complex Care Needs
MeSH Terms: conditions — Gastrointestinal Neoplasms; Ovarian Neoplasms; Ascites

STUDY DESIGN:
Intervention Model Description: Phase I: Single-arm study with up to 20 ovarian cancer patients and their informal caregivers run-in.
  Phase II: Two-arm pilot RCT with 60 gynecologic or gastrointestinal cancer patients and their informal caregivers (30 dyads in each arm).
Who Masked: Outcomes Assessor
Masking Description: Clinical research assistant blinded to randomized study arms; will conduct structured interview at baseline, prior to randomization, and 4 weeks post randomization +/- 2 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bolster (Experimental): * Bolster provides participants with longitudinal nursing support across care settings,
  * A smartphone-based symptom management app,
  * A print and web-based symptom management toolkit,
  * Advance care planning to ensure that the patient receives care that is congruent with her informed preferences
  * BOLSTER includes a total of 6 contacts with a study nurse over 4 weeks
  * Daily contact via a smartphone-based symptom app which queries patients about their symptoms using questions from the PRO-CTCAE, risk-stratifies their symptoms, and provides tailored symptom management advice
  Interventions: Behavioral: BOLSTER
- Enhanced Discharge Planning (EDP) (Other): * Medication education,
  * Self-management strategies for symptoms,
  * Skills training,
  * A list of red flag symptoms and numbers for who to call
  Interventions: Other: Enhanced Discharge Planning (EDP)

INTERVENTIONS:
Behavioral: BOLSTER — BOLSTER provides patients and caregivers with education and skills training, symptom management, and support across care settings over a four-week period.
  Arms: Bolster
Other: Enhanced Discharge Planning (EDP) — EDP provides patients and caregivers a single session of education and skills training, symptom management, and support.
  Arms: Enhanced Discharge Planning (EDP)

SUMMARY:
This research study is evaluating a new intervention, BOLSTER, which was designed to provide more support for patients with gynecologic and gastrointestinal cancers and their caregivers after a hospitalization.

DETAILED DESCRIPTION:
Hospitalizations can be difficult for patients with cancer, especially when they are transitioning home. Patients and caregivers are often expected to perform complex medical and nursing tasks with little or no preparation. Patients and caregivers report high levels of unmet needs for information about how best to manage symptoms and new medical procedures (such as managing new tubes, lines or drains).

The study team has developed a research project which aims to address these needs. If a patient agrees to participate in the study, she will take part in a program called BOLSTER (Building Out Lifelines for Safety, Trust, Empowerment and Renewal). BOLSTER will provide patients and caregivers with education and skills training, symptom management, and support across care settings.

ELIGIBILITY:
Patient inclusion criteria

* Adults (≥18 years old);
* GYN or GI cancers receiving anti-neoplastic therapy;
* Hospitalized, recently hospitalized (i.e. within the first 2 visits after a hospitalization), or recent outpatient placement of tube, line, or drain (e.g. PleurX catheter);
* Plan to receive ongoing care at DFCI;
* Willingness to be audio taped for the study (for monitoring of study fidelity).
* Have complex care needs (e.g. an ostomy, ileostomy, a gastric tube, percutaneous nephrostomy tubes, a PleurX catheter, or need for total parenteral nutrition)

Patient exclusion criteria

* Unable to read and respond to questions in English;
* Cognitive impairment;
* Unable to complete the baseline interview;
* Plan for immediate hospice referral

Caregiver inclusion criteria

* Adults (≥18 years old);
* Family member or friend of an eligible patient;
* Willingness to be audio taped for the study (for monitoring of study fidelity);
* Willingness to participate in study visits

Caregiver exclusion criteria:

* Unable to read and respond to questions in English,
* Cognitive impairment
* Unable to complete the baseline interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexi A Wright, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- 25873, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pozzar RA, Enzinger AC, Poort H, Furey A, Donovan H, Orechia M, Thompson E, Tavormina A, Fenton ATHR, Jaung T, Braun IM, DeMarsh A, Cooley ME, Wright AA. Developing and Field Testing BOLSTER: A Nurse-Led Care Management Intervention to Support Patients and Caregivers following Hospitalization for Gynecologic Cancer-Associated Peritoneal Carcinomatosis. J Palliat Med. 2022 Sep;25(9):1367-1375. doi: 10.1089/jpm.2021.0618. Epub 2022 Mar 17. PMID 35297744
- [Derived] Pozzar RA, Enzinger AC, Howard C, Tavormina A, Matulonis UA, Campos S, Liu JF, Horowitz N, Konstantinopoulos PA, Krasner C, Wall JA, Sciacca K, Meyer LA, Lindvall C, Wright AA. Feasibility and acceptability of a nurse-led telehealth intervention (BOLSTER) to support patients with peritoneal carcinomatosis and their caregivers: A pilot randomized clinical trial. Gynecol Oncol. 2024 Sep;188:1-7. doi: 10.1016/j.ygyno.2024.06.001. Epub 2024 Jun 7. PMID 38851039

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase Ia: 10-week Pre-pilot Patients; Phase Ia: 10-week Pre-pilot Caregivers: In this single arm pre-pilot, patients and caregiver dyads were offered a total of 12 contacts with a BOLSTER study nurse over 10 weeks and daily contact via a smartphone-based symptom app which queries patients about their symptoms using questions from the PRO-CTCAE, risk-stratifies their symptoms, and provides tailored symptom management advice. Participants also had access to web-based symptom management and medical skills training.
- Phase Ib: 4-week Pre-pilot Patients; Phase Ib: 4-week Pre-pilot Caregivers: The second, abbreviated iteration of the intervention consisted of a single arm pre-pilot, in which patient and caregiver dyads were offered a total of 6 contacts with a BOLSTER study nurse over 4 weeks and daily contact via a smartphone-based symptom app which queries patients about their symptoms using questions from the PRO-CTCAE, risk-stratifies their symptoms, and provides tailored symptom management advice. Participants also had access to web-based symptom management and medical skills training.
- Phase II (RCT): BOLSTER Arm Patients; Phase II (RCT): BOLSTER Arm Caregivers: BOLSTER provides participants with longitudinal nursing support across care settings, a smartphone-based symptom management app, a print and web-based symptom management toolkit, and advance care planning to ensure that the patient receives care that is congruent with her informed preferences. BOLSTER includes a total of 6 contacts with a study nurse over 4 weeks. Daily contact via a smartphone-based symptom app which queries patients about their symptoms using questions from the PRO-CTCAE, risk-stratifies their symptoms, and provides tailored symptom management advice.
- Phase II (RCT): EDP Arm Patients; Phase II (RCT): EDP Arm Caregivers: Enhanced Discharge Planning (EDP): EDP provides patients and caregivers a single session of education and skills training, symptom management, and support. The EDP participants received medication education, self-management strategies for symptoms, skills training, and a list of red flag symptoms and numbers for who to call.
Period: Overall Study
Arm/Group | Phase Ia: 10-week Pre-pilot Patients | Phase Ia: 10-week Pre-pilot Caregivers | Phase Ib: 4-week Pre-pilot Patients | Phase Ib: 4-week Pre-pilot Caregivers | Phase II (RCT): BOLSTER Arm Patients | Phase II (RCT): BOLSTER Arm Caregivers | Phase II (RCT): EDP Arm Patients | Phase II (RCT): EDP Arm Caregivers
Started | 6 | 6 | 5 | 4 | 29 | 17 | 32 | 22
Completed | 3 | 3 | 5 | 4 | 21 | 11 | 20 | 15
Not Completed | 3 | 3 | 0 | 0 | 8 | 6 | 12 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase Ia: 10-week Pre-pilot Patients | Phase Ia: 10-week Pre-pilot Caregivers | Phase Ib: 4-week Pre-pilot Patients | Phase Ib: 4-week Pre-pilot Caregivers | Phase II (RCT): BOLSTER Arm Patients | Phase II (RCT): BOLSTER Arm Caregivers | Phase II (RCT): EDP Arm Patients | Phase II (RCT): EDP Arm Caregivers | Total
Number analyzed (Participants) | 6 | 6 | 5 | 4 | 29 | 17 | 32 | 22 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (7.31) | 64 (6.63) | 58 (14.03) | 62 (12.48) | 60 (10.17) | 59 (9.54) | 62 (7.51) | 60 (10.21) | 61 (9.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 5 | 1 | 25 | 10 | 31 | 7 | 86
  Male | 0 | 5 | 0 | 3 | 4 | 7 | 1 | 15 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 5
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 5
  Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
  White | 6 | 6 | 4 | 3 | 24 | 14 | 26 | 20 | 103
  Other | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 4
  I don't know/refuse to answer | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Ethnicity [Count of Participants; unit: Participants]
  Hispanic or LatinX | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 4
  Not Hispanic or LatinX | 6 | 6 | 5 | 4 | 27 | 16 | 27 | 21 | 112
  Missing | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 5
Marital Status [Count of Participants; unit: Participants]
  Married | 5 | 6 | 5 | 4 | 22 | 16 | 26 | 20 | 104
  Divorced/Separated | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 6
  Single, never married | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 5
  Widowed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Partnered | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3
  I don't know/refused | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Highest Level of Education [Count of Participants; unit: Participants]
  8th grade or less | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  9 - 11th grade | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
  High school graduate / GED | 1 | 2 | 0 | 1 | 1 | 2 | 3 | 1 | 11
  Vocational / Technical training | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 4
  Associate degree / some college | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 3 | 8
  Bachelor's degree | 2 | 1 | 3 | 2 | 11 | 3 | 11 | 8 | 41
  Advanced degree | 2 | 3 | 0 | 1 | 14 | 11 | 14 | 7 | 52
  Refuse to answer | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the BOLSTER Intervention
Description: ≥50% consent-to-approach ratio
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Groups:
- Patients Approached: The number of patients that study staff approached regarding participation in the study
Arm/Group | Patients Approached
Number analyzed (Participants) | 95
Participants
  Consented | 73
  Did not consent | 22

2. Secondary Outcome: Acceptability of the BOLSTER Intervention
Description: ≥70% participants "agree" or "strongly agree" that they would recommend BOLSTER to other patients; and ≥70% participants "agreed or "strongly agreed" that they were satisfied with the BOLSTER intervention. Note that this measure only includes data from the RCT portion of the study, as the Phases 1a and 1b were designed to refine the intervention.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II (RCT): BOLSTER Arm Patients | Phase II (RCT): BOLSTER Arm Caregivers
Number analyzed (Participants) | 22 | 10
Participants
  Acceptability - "I have been satisfied with the BOLSTER program sessions...": Strongly agree | 14 | 8
  Acceptability - "I have been satisfied with the BOLSTER program sessions...": Agree | 6 | 2
  Acceptability - "I have been satisfied with the BOLSTER program sessions...": Neither agree nor disagree | 2 | 0
  Acceptability - "I would recommend the BOLSTER program to other patients...": Strongly agree | 16 | 8
  Acceptability - "I would recommend the BOLSTER program to other patients...": Agree | 5 | 2
  Acceptability - "I would recommend the BOLSTER program to other patients...": Neither agree nor disagree | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 2 months while patients were on study, since this is a minimal risk study.
Arm/Group | Phase Ia: 10-week Pre-pilot Patients | Phase Ia: 10-week Pre-pilot Caregivers | Phase Ib: 4-week Pre-pilot Patients | Phase Ib: 4-week Pre-pilot Caregivers | Phase II (RCT): BOLSTER Arm Patients | Phase II (RCT): BOLSTER Arm Caregivers | Phase II (RCT): EDP Arm Patients | Phase II (RCT): EDP Arm Caregivers
All-Cause Mortality (participants affected / at risk) | 3/6 | 0/6 | 0/5 | 0/4 | 5/29 | 0/17 | 3/32 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/5 | 0/4 | 0/29 | 0/17 | 0/32 | 0/22
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/5 | 0/4 | 0/29 | 0/17 | 0/32 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/47/NCT03367247/Prot_SAP_000.pdf